CLINICAL TRIAL: NCT04688190
Title: Choice of Optimal Transcatheter Treatment for Mitral Insufficiency Registry
Acronym: CHOICE-MI
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Montreal Heart Institute (Other); University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Sebastian Ludwig, Sebastian Ludwig, M.D., Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: CHOICE-MI
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Transcatheter Mitral Valve Implantation (TMVI): Patients with successful TMVI screening, who underwent Transcatheter Mitral Valve Implantation subsequently. All devices may be included.
- Interventional mitral valve edge-to-edge repair (E2E): Patients with TMVI screening failure, who subsequently underwent interventional mitral valve edge-to-edge repair.
- Mitral valve surgery (Surgery): Patients with TMVI screening failure, who subsequently underwent mitral valve surgery (i.e., mitral valve repair or replacement).
- Medical therapy (OMT): Patients with TMVI screening failure, who subsequently underwent conservative or optimal medical therapy (OMT).

SUMMARY:
This multinational, investigator-initiated, retrospective study aims to investigate outcomes of patients, who underwent transcatheter mitral valve implantation (TMVI), in comparison to those screened for TMVI but deemed ineligible, who subsequently underwent interventional mitral valve edge-to-edge repair, mitral valve surgery or medical/conservative therapy.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant mitral insufficiency
* patient underwent screening for TMVI
* echocardiography data at baseline (and after TMVI, E2E and surgery)
* follow-up of at least 30 days

Exclusion Criteria:

- age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aimes to include all patients with significant mitral insufficiency, who underwent screening for possible transcatheter mitral valve implantation (TMVI), irrespective of the subsequent therapy.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitral insufficiency grade 2+ or more | 12 months
  Mitral insufficiency measured by transthoracic echocardiography. Assessment of MI severity according to current guidelines (ESC/EACTS and ACC/AHA) for valvular heart disease.
Freedom from device-related complications | 30 days

SECONDARY OUTCOMES:
Combined all-cause mortality or rehospitalization for congestive heart failure | 12 months
All-cause mortality | 12 months
Cardiovascular mortality | 12 months
Rehospitalization for congestive heart failure | 12 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization, e.g. as assessed by patient interviews.
Combined cardiovascular mortality or rehospitalization for congestive heart failure | 12 months
Unplanned mitral valve intervention | 12 months
  Incidence of unplanned surgical or transcatheter re-intervention, heart transplantation or left ventricular assist device implantation, e.g. as assessed by patient interviews.
Combined all-cause mortality, rehospitalization for congestive heart failure or unplanned mitral valve intervention | 12 months
Combined cardiovascular mortality, rehospitalization for congestive heart failure or unplanned mitral valve intervention | 12 months
New York Heart Association (NYHA) stage III or IV | 12 months
  Assessment of New York Heart Association (NYHA) classification stage (in- or outpatient) after 12 months follow-up, as assessed by patient interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Conradi, MD, Principal Investigator — University Heart and Vascular Center Hamburg; Thomas Modine, MD, Principal Investigator — University Hospital, Bordeaux; Sebastian Ludwig, MD, Principal Investigator — University Heart and Vascular Center Hamburg; Walid Ben Ali, MD, Principal Investigator — Montreal Heart Institute; Alison Duncan, MD, Principal Investigator — Royal Brompton Hospital, London; Gilbert Tang, MD, Principal Investigator — Mount Sinai Medical Center, NYC; Juan F Granada, MD, Principal Investigator — Cardiovascular Research Foundation, New York, USA
Locations (26):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Houston Methodist Hospital, Houston, Texas
- St Vincent's Hospital, Sydney, Australia
- Canada (2):
  - Toronto Heart Center, Toronto
  - St. Paul's Hospital, Vancouver
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - CHU Bordeaux, Bourdeaux
  - Lille University Hospital, Lille
  - Civils Hospices of Lyon, Lyon
  - Clinique Pasteur, Toulouse
- Germany (9):
  - HDZ Bad Oeynhausen, Bad Oeynhausen
  - German Heart Center Berlin, Berlin
  - Heart Center Bonn, Bonn
  - University Hospital of Cologne, Cologne
  - Goethe-Universität - University Hospital Frankfurt, Frankfurt
  - University Heart and Vascular Center Hamburg, Hamburg
  - Heart Center of the University Medical Center Mainz, Mainz
  - German Heart Centre Munich, Munich
  - LMU Munich, Munich
- San Raffaele University Hospital, Milan, Italy
- Rikshospitalet, Oslo University Hospital (OUS), Oslo, Norway
- Switzerland (2):
  - Inselspital Bern, Bern
  - USZ Zurich, Zurich
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - St Thomas' Hospital - London, London

REFERENCES:
- [Derived] Ludwig S, Coisne A, Hamzi K, Ben Ali W, Scotti A, Koell B, Duncan A, Makkar R, Akodad M, Bleiziffer S, Nickenig G, Kaneko T, Ruge H, Adam M, Sondergaard L, Dahle G, Taramasso M, Walther T, Kempfert J, Obadia JF, Chehab O, Tang GHL, Goel S, Fam N, Denti P, Praz F, von Bardeleben RS, Hausleiter J, Latib A, Conradi L, Modine T, Pezel T, Granada JF; CHOICE-MI Investigators. Phenotypic clustering analysis of patients rejected for mitral valve interventions: implications for future transcatheter technologies. Eur Heart J Cardiovasc Imaging. 2025 Jul 31;26(8):1452-1463. doi: 10.1093/ehjci/jeaf141. PMID 40329826
- [Derived] Coisne A, Ludwig S, Scotti A, Ben Ali W, Weimann J, Duncan A, Webb JG, Kalbacher D, Rudolph TK, Nickenig G, Hausleiter J, Ruge H, Adam M, Petronio AS, Dumonteil N, Sondergaard L, Adamo M, Regazzoli D, Garatti A, Schmidt T, Dahle G, Taramasso M, Walther T, Kempfert J, Obadia JF, Redwood S, Tang GHL, Goel S, Fam N, Metra M, Andreas M, Muller DW, Denti P, Praz F, von Bardeleben RS, Leroux L, Latib A, Granada JF, Conradi L, Modine T; CHOICE-MI Investigators. Outcomes Following Transcatheter Mitral Valve Replacement Using Dedicated Devices in Patients With Mitral Annular Calcification. JACC Cardiovasc Interv. 2024 Sep 23;17(18):2141-2153. doi: 10.1016/j.jcin.2024.07.038. Epub 2024 Sep 4. PMID 39243262
- [Derived] Ludwig S, Conradi L, Cohen DJ, Coisne A, Scotti A, Abraham WT, Ben Ali W, Zhou Z, Li Y, Kar S, Duncan A, Lim DS, Adamo M, Redfors B, Muller DWM, Webb JG, Petronio AS, Ruge H, Nickenig G, Sondergaard L, Adam M, Regazzoli D, Garatti A, Schmidt T, Andreas M, Dahle G, Walther T, Kempfert J, Tang GHL, Redwood S, Taramasso M, Praz F, Fam N, Dumonteil N, Obadia JF, von Bardeleben RS, Rudolph TK, Reardon MJ, Metra M, Denti P, Mack MJ, Hausleiter J, Asch FM, Latib A, Lindenfeld J, Modine T, Stone GW, Granada JF; CHOICE-MI and the COAPT Trial Investigators. Transcatheter Mitral Valve Replacement Versus Medical Therapy for Secondary Mitral Regurgitation: A Propensity Score-Matched Comparison. Circ Cardiovasc Interv. 2023 Jun;16(6):e013045. doi: 10.1161/CIRCINTERVENTIONS.123.013045. Epub 2023 May 16. PMID 37194288